CLINICAL TRIAL: NCT02520037
Title: Fluid Responsiveness Prediction Using Extra Systoles in Critically Ill Patients
Brief Title: Fluid Responsiveness Prediction Using Extra Systoles
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: University of Aarhus
Record Dates: First submitted 2015-08-03; First posted 2015-08-11 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-05

CONDITIONS: Fluid Responsiveness
Keywords: Fluid responsiveness; Volume responsiveness; Hemodynamics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Fluids are generally administered to patients in order to improve circulation. However, fluids do not always improve circulation and fluids have side effects. Unfortunately, it is difficult to predict whether fluid administration improves the circulation, i.e. it is difficult to predict fluid responsiveness The overall aim of this observational study is to investigate if analysis of spontaneously occuring extra systoles can give the answer: The second beat in the extra systole - the post ectopic beat - is a normal sinus beat but it has experienced the compensatory pause, i.e. this beat is associated with increased filling time and in turn associated with increased filling. As such, the post ectopic beat shows how the heart responds to increased filling. Therefore, the hypothesis of this study is that the hemodynamic response to the increased filling at the post ectopic beat (compared with sinus beats) can predict fluid responsiveness

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a 500 ml volume expansion
* Patients without atrial fibrillation
* Patients equipped with ECG, arterial pressure and non-invasive cardiac output monitoring

Exclusion Criteria:

* Changes in anesthetic, vasoactive or inotropic drugs during the study period (30 minutes before fluid infusion initiation to end of fluid infusion).
* Changes in positive end-expiratory pressure the study period
* Changes in bed positioning the study period
* Infusion time with crystalloids exceeding 30 minutes
* Infusion time with colloids exceeding 75 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to a University Hospital intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Change in stroke volume (SV) following fluid administration. A positive fluid response is defined as a 15% or more increase in SV | Change in SV from immediately before fluid infusion (t=0 min) to immediately after fluid administration (t < 30 min for crystalloid infusions; t < 75 min for colloid infusions)
  A positive fluid response is defined as a 15% or more increase in SV. From the arterial pressure curve, post ectopic changes (comparing with 10 preceding sinus beats) in systolic blood pressure and pre-ejection period will be derived and used to predict the fluid response. Time frame used is the 30 minutes prior to the volume expansion (from t = -30 min to t = 0 min)

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus C, Denmark